CLINICAL TRIAL: NCT01056549
Title: Exenatide (Byetta ®) Regulation of Intestinal and Hepatic Lipoprotein Particle Production in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Gary Lewis, Professor, Department of Medicine and Physiology, University Health Network, Toronto
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: REB 09-0428-B
Record Dates: First submitted 2009-11-12; First posted 2010-01-26 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Hyperlipidemia
Keywords: Intestinal lipoprotein; Apo B48 and apoB100; Pancreatic clamp; GLP-1 agonist
MeSH Terms: conditions — Hyperlipidemias | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- exenatide subcutaneous injection (Experimental): Study A: lipoprotein turnover following subcutaneous exenatide administration, under conditions of pancreatic clamp. Study B: lipoprotein turnover study following subcutaneous placebo administration, under conditions of pancreatic clamp.
  Interventions: Drug: exenatide

INTERVENTIONS:
Drug: exenatide — In each study, the subjects will receive s.c. injection of either exenatide or matched placebo, in the Metabolic Testing Center and 2 hours prior to the start of the lipoprotein turnover study. Subjects will be blinded with regard to the treatments.
  Other Names: Byetta

SUMMARY:
Exenatide acutely inhibits intestinal lipoprotein particle production. We are unable to speculate whether exenatide affects hepatic lipoprotein production in humans since there is currently no evidence from animal models or in vitro studies that have demonstrated an effect

DETAILED DESCRIPTION:
Subjects will receive an infusion of stable isotope enriched acetate, leucine and a bolus of glycerol in order to measure the rates of fatty acid synthesis, apolipoprotein and triglyceride turnover respectively. This in vivo stable isotope enrichment methodology has been widely established and used by investigators around the world for more than 30 years to examine the metabolism of various metabolites in humans.

Following an overnight fast, at approximately 9am on day 1 of the study the subject will be admitted to hospital and will have a 30ml fasting blood sample drawn for analysis of plasma glucose, total plasma cholesterol, LDL-cholesterol, HDL cholesterol, triglycerides (TG), free fatty acids (FFA), insulin, GLP-1, growth hormone, glucagon, stable isotope enrichment and a more detailed analysis of triglyceride rich lipoprotein (TRL) composition (lipid and apolipoprotein content). A radio-opaque polyvinyl feeding tube (Entriflex NG Tube 55'' [140cm] 10fr Item # 8884721055, Kendall Products, Tyco Healthcare, Toronto, ON) will be inserted through the nose into the stomach, with enough length provided for migration of the tip into the duodenum. The subject will be administered 10 mg metoclopramide orally to facilitate transport of the tip of the tube into the duodenum. The subject will be allowed to eat regular meals during the day but will fast overnight after 7pm and will remain fasting for the duration of the study. Water ad lib will be allowed. At approximately 3pm on day 1 an abdominal X-Ray will confirm the position of the tube in the duodenum. At 4pm 2 iv's will be inserted into a superficial vein in each forearm, one for infusion and one for sampling. An infusion of 1-13C acetate (15 gm in a bag of ½ N saline at 32ml/hr) will begin after the iv's have been inserted and will be infused for the remainder of the study, which is 27 hours.

Starting at 4am a synthetic triglyceride emulsion, Intralipid (20% solution, Baxter Canada) , will be infused through the feeding tube into the duodenum at a rate of 40 ml/hr for the duration of the experiment (ie until 7pm that evening). This will provide a steady state fed state for the subsequent assessment of lipoprotein turnover kinetics.

The subjects will receive, in random order, either exenatide 10 mg or equivalent volume of saline subcutaneously at 7am on day 2 of the hospitalization (i.e. at -2hr) during the first of the two studies. The pancreatic clamp will begin at 7am (-2hr), immediately following administration of either exenatide or saline and continue throughout the subsequent 12 hours (until 7pm). . During the pancreatic clamp the subjects will receive an iv infusion of glucagon (0.65ng/kg/min), growth hormone (Humatrope, 3.0 ng/kg/min), somatostatin (sandostatin, 25 µg/hr) and insulin (Novolin R, 0.05 mU/kg/min).

At 9 am (we will refer to this time point as 0hr of the lipoprotein turnover study), the lipoprotein turnover study will begin. An iv bolus of deuterated-glycerol (d5-glycerol, 75 mmol/kg) will be administered, followed by a primed-constant infusion of deuterated leucine; d3-leucine, (10 mmol/kg bolus followed by 10 mmol/kg/hr for 10 hours). Blood samples will be collected prior to and at regular time intervals for 10 hours after the iv bolus of d3-glycerol and start of the constant infusion of d3-leucine (for assessment of lipoprotein kinetics). Blood samples will be collected prior to (30ml at -2hr, 10ml at -1hr and 30ml at 0hr) and 5min and 15min (10ml each) and then 30ml each at 30min, 1hr, 2hr, 3hr, 4hr, 5hr, 6hr (only 10ml),7hr, 8hr, 9hr and 10hr after administration of d5-glycerol and start of d3-leucine infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20 kg/m2 to 25 kg/m2
3. Hemoglobin above 130g/L.
4. Normal glucose tolerance in response to a 75g, 2-hr OGTT

Exclusion Criteria:

1. Subject has a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (Cr > 1.5 mg/dL), genitourinary, hematological systems, or has severe uncontrolled treated or untreated hypertension (sitting diastolic BP > 100 or systolic > 180) or proliferative retinopathy
3. History of diabetes or OGTT indicative of diabetes or impaired glucose tolerance.
4. Any history of a MI or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on ECG, unstable angina, or decompensated heart failure.
5. Any laboratory values: AST > 2x ULN; ALT > 2x ULN TSH > 6 mU/l
6. Current addiction to alcohol or substances of abuse as determined by the investigator.
7. Mental incapacity, unwillingness or language barrier precluding adequate understanding or cooperation
8. Taking any prescription or non-prescription medications at the time of the study
9. Having donated blood three months prior to and three months post study procedures
10. A pregnancy test will be performed 1 to 3 days prior to each study in all female subjects. Those who test positive for pregnancy will be excluded.
11. No clinical evidence of neoplasms which have been known to overexpress GLP-1 receptors i.e. pheochromocytomas, brain tumors and embryonic tumors.
12. Hypersensitivity to egg-, soya-,or peanut protein or previous allergy to intralipid
13. Those with known sensitivity to metoclopramide

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The objective is to examine the change in apoB48 production rate after one subcutaneous injection of exenatide, under conditions of a pancreatic clamp and a steady state fed state. | over 10 hours

SECONDARY OUTCOMES:
The secondary objective is to examine the change in apoB100 production rate in the same conditions, and the secondary measure is the difference between exenatide and placebo in the mean production of TRL-apoB100 | over 10 hours

CONTACTS AND LOCATIONS:
Overall Officials: gary F Lewis, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Xiao C, Bandsma RH, Dash S, Szeto L, Lewis GF. Exenatide, a glucagon-like peptide-1 receptor agonist, acutely inhibits intestinal lipoprotein production in healthy humans. Arterioscler Thromb Vasc Biol. 2012 Jun;32(6):1513-9. doi: 10.1161/ATVBAHA.112.246207. Epub 2012 Apr 5. PMID 22492091